CLINICAL TRIAL: NCT00073320
Title: Pharmacokinetics, Tolerability, and Safety of Paliperidone After Repeated Intramuscular Injection of Paliperidone Palmitate in the Arm or the Buttock of Subjects With Schizophrenia
Brief Title: Intramuscular Injections of Paliperidone Palmitate in the Arm or Buttock of Subjects With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR004462
Record Dates: First submitted 2003-11-19; First posted 2003-11-21 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2010-04

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Paliperidone palmitate; R092670; antipsychotic
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate

INTERVENTIONS:
Drug: Paliperidone Palmitate

SUMMARY:
The purpose of the study is to compare the pharmacokinetic parameters (blood concentrations) of i.m. paliperidone palmitate after administration in 2 different injection sites (deltoid or gluteal).

DETAILED DESCRIPTION:
An i.m. paliperidone palmitate long-acting formulation is under development with the aim to provide a sustained and stable level of paliperidone during each treatment cycle. The goal of this study is to determine the similarity in pharmacokinetic (blood levels) and safety profile after 2 intramuscular injections of paliperidone palmitate in the arm (deltoid muscle) and the buttock (gluteal muscle), in the dose range that will be covered in later Phase 3 trials (25 - 150 mg eq.). This is a repeated-dose, open-label, parallel group study in patients with schizophrenia. The study consists of an up to 5-day screening period, an up to 3-day tolerability period, a 14-day washout period, and a 64-day treatment period. As paliperidone is the active metabolite of risperidone, all patients will be exposed to oral risperidone during the screening period to confirm that they do not develop allergic reactions to risperidone, and to help the investigator to assign patients to 1 of the 2 treatment doses. There will be a washout of at least 2 weeks after the last oral risperidone intake before patients receive the first injection of paliperidone palmitate. Each treatment group (arm or buttock injection) will receive 2 consecutive i.m. injections of the long-acting formulation of paliperidone palmitate with a one-week interval. Whole blood samples will be collected for the determination of paliperidone palmitate and paliperidone concentrations in plasma. Whole blood samples will be obtained by venipuncture (needle stick) immediately before (pre-dose) and at 4, 8, 12, 24, 48, 72, and 96 hours after the 1st and 2nd injections of paliperidone palmitate. Following the collection of the 96-hour blood sample after the 2nd injection, additional samples will be collected every 3 to 7 days through the end of the 64-day treatment period. Safety will assessed throughout the study by monitoring adverse events; changes in clinical laboratory results; tardive dyskinesia will be rated using the Abnormal Involuntary Movement Scale (AIMS), akathisia will be rated according to the Barnes Akathisia Rating Scale (BARS), extrapyramidal symptoms will be evaluated using the Simpson-Angus Rating Scale (SAS); physical examinations; electrocardiograms (ECGs); and patient evaluation of the injection site. Paliperidone palmitate (25 or 150 mg eq.), 2 i.m. doses administered at a 1-week interval. Depending on the randomized treatment group, each patient will receive 3 doses of oral risperidone: either 1 mg once daily for 3 days or 2 mg once on the 1st day, 4 mg once on the 2nd day, and 6 mg once on the 3rd day.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of schizophrenia
* clinically stable with no change in current antipsychotic medications
* meet PANSS score criteria
* have a body mass index (BMI) between 15 and 35 kilogram (kg)/meter (m)2.

Exclusion Criteria:

* Patients with DSM-IV diagnosis of alcohol or substance dependence, with the exception of nicotine or caffeine dependence
* involuntarily-committed
* have moderately severe or severe EPS symptoms
* history of malignant neuroleptic syndrome
* have current suicidal ideation or demonstrates violence
* current presence of any significant or unstable medication condition
* treatment with any protocol disallowed therapies
* clinically significant result from screening laboratory or ECG.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2003-08; Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
To explore the comparability of pharmacokinetic parameter estimates of paliperidone and paliperidone palmitate between the 2 injection sites.

SECONDARY OUTCOMES:
Incidence of adverse events, labs and ECGs throughout study.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.